CLINICAL TRIAL: NCT01895218
Title: A, Randomized Comparative, Open-Label Study of Intravenous Iron Isomaltoside 1000 (Monofer®) Administered by High Single Dose In-fusions or Standard Medical Care in Women After Postpartum Haemorrhage
Brief Title: Treatment of Women After Postpartum Haemorrhage
Acronym: PP-01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Collaborators: BioStata (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PP-01
Record Dates: First submitted 2013-06-26; First posted 2013-07-10 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Postpartum Haemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — iron isomaltoside 1000

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iron isomaltoside 1000 (Monofer®) (Experimental)
  Interventions: Drug: Iron isomaltoside 1000
- Standard medical Care (Active Comparator)
  Interventions: Other: Standard medical Care

INTERVENTIONS:
Drug: Iron isomaltoside 1000 — A single dose of 1200 mg iron isomaltoside 1000 is given. The dose is diluted in 100 ml 0.9 % sodium chloride and given over approximately 15 min.
  Other Names: Monofer®
  Arms: Iron isomaltoside 1000 (Monofer®)
Other: Standard medical Care — Standard medical Care is most often to recommend women with PPH to continue oral iron supplementation as recommended during pregnancy or to advise the subject to take 100 mg oral iron 1-2 times a day
  Arms: Standard medical Care

SUMMARY:
The primary purpose of this study is to compare the efficacy of IV high single dose infusion of iron isomaltoside 1000 to standard medical care in women with PPH evaluated as physical fatigue.

ELIGIBILITY:
Inclusion Criteria:

1. Women with PPH ≥ 700 and ≤ 1000 mL or PPH > 1000 mL and Hb > 6.5 g/dL (4.0 mmol/L) measured > 12 hours after delivery
2. Willingness to participate and signed the informed consent form

Exclusion Criteria:

1. Women aged < 18 years
2. Multiple births
3. Peripartum RBC transfusion
4. Known iron overload or disturbances in utilisation of iron (e.g. haemochromatosis and haemosiderosis)
5. Known hypersensitivity to parenteral iron or any excipients in the investigational drug products
6. Women with a history of active asthma within the last 5 years or a history of multiple allergies
7. Known decompensated liver cirrhosis and active hepatitis
8. Women with HELLP (Haemolysis Elevated Liver enzymes Low Platelet count) syndrome (defined according to "Dansk Selskab for Obstetrik og Gynækologi guidelines")
9. Active acute infection assessed by clinical judgement
10. Rheumatoid arthritis with symptoms or signs of active joint inflammation
11. History of anaemia caused by e. g. thalassemia, hypersplenism or haemolytic anaemia (known haematologic disorder other than iron deficiency)
12. Not able to read, speak and understand the Danish language
13. Participation in any other clinical study where the study drug has not passed 5 half-lives prior to the baseline
14. Any other medical condition that, in the opinion of the Investigator, may cause the patient to be unsuitable for completion of the study or place the patient at potential risk from being in the study. For example, a malignancy, uncontrolled hypertension, unstable ischaemic heart disease or uncontrolled diabetes mellitus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Physical fatigue | From exposure to 12 weeks post-exposure
  The primary objective of this study is to compare efficacy of IV high single dose infusion of iron isomaltoside 1000 to standard medical care in women with PPH evaluated as physical fatigue.

SECONDARY OUTCOMES:
Change in Hb concentration | From exposure to week 1, 3, 8 and 12 post-exposure
Change in concentrations of p-ferritin | From exposure to day 3, week 1, 3, 8 and 12 post-exposure
Change in Fatigue symptoms | From exposure to day 3, week 1, 3, 8 and 12 post-exposure
Change in postpartum depression symptoms | From exposure to 12 weeks post-exposure
Breastfeeding | From exposure to 12 weeks post-exposure
RCB transfusions | From exposure to 12 weeks post-exposure
Adverse drug reactions (ADRs) | From exposure to day 3, week 1, 3, 8 and 12 post-exposure
Change in concentrations of p-iron | From exposure to day 3, week 1, 3, 8 and 12 post-exposure
Change in concentrations of p-transferrin | From exposure to day 3, week 1, 3, 8 and 12 post-exposure
Change in concentrations of transferrin saturation (TSAT) | From exposure to day 3, week 1, 3, 8 and 12 post-exposure
Change in concentrations of reticulocyte count | From exposure to day 3, week 1, 3, 8 and 12 post-exposure
Change in concentrations of mean reticulocyte haemoglobin content (CHr) | From exposure to day 3, week 1, 3, 8 and 12 post-exposure
Change in haematology parameters | From exposure to day 3, week 1, 3, 8 and 12 post-exposure

OTHER OUTCOMES:
Change in anaemia symptoms | From exposure to day 3, week 1, 3, 8 and 12 post-exposure
Change in gastrointestinal symptoms | From exposure to day 3, week 1, 3, 8 and 12 post-exposure

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen, Denmark

REFERENCES:
- [Derived] Holm C, Thomsen LL, Langhoff-Roos J. Intravenous iron isomaltoside treatment of women suffering from severe fatigue after postpartum hemorrhage. J Matern Fetal Neonatal Med. 2019 Sep;32(17):2797-2804. doi: 10.1080/14767058.2018.1449205. Epub 2018 Mar 20. PMID 29558233
- [Derived] Holm C, Thomsen LL, Norgaard A, Langhoff-Roos J. Intravenous iron isomaltoside 1000 administered by high single-dose infusions or standard medical care for the treatment of fatigue in women after postpartum haemorrhage: study protocol for a randomised controlled trial. Trials. 2015 Jan 14;16:5. doi: 10.1186/1745-6215-16-5. PMID 25588587